CLINICAL TRIAL: NCT03437733
Title: Multi-electrode Radiofrequency Balloon Catheter Use for the Isolation of the Pulmonary Veins.
Acronym: SHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI_2017_01
Record Dates: First submitted 2018-02-13; First posted 2018-02-19 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Radiofrequency Ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Experimental): Ablation with Multi-electrode Radiofrequency (RF) Balloon Catheter
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Device: Radiofrequency Ablation — RF ablation using multi-electrode radiofrequency balloon catheter and multi-electrode circular diagnostic catheter

SUMMARY:
This clinical investigation is a prospective, multicenter, single arm clinical evaluation utilizing the multi-electrode radiofrequency balloon catheter and the multi-electrode circular diagnostic catheter.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to assess the safety and acute effectiveness of the multi-electrode radiofrequency balloon catheter and multi-electrode circular diagnostic catheter when used for the isolation of the pulmonary veins in the treatment of Paroxysmal Atrial Fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Symptomatic Paroxysmal AF.
2. Selected for atrial fibrillation (AF) ablation procedure for pulmonary vein isolation.
3. Able and willing to comply with uninterrupted per-protocol anticoagulation requirements
4. Age 18-75 years.
5. Able and willing to comply with all pre-, post- and follow-up testing and requirements.
6. Signed Patient Informed Consent Form.

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Previous surgical or catheter ablation for AF.
3. Anticipated to receive ablation outside the PV ostia and Cavo-triscuspid-isthmus (CTI) region
4. Previously diagnosed with persistent, longstanding AF and/or continuous AF > 7 days, or > 48 hrs terminated by cardioversion.
5. Any percutaneous coronary intervention (PCI) within the past 2 months.
6. Valve repair or replacement and presence of a prosthetic valve.
7. Any carotid stenting or endarterectomy.
8. Coronary artery bypass grafting (CABG), cardiac surgery (e.g. ventriculotomy, atriotomy), or valvular cardiac surgical or percutaneous procedure within the past 6 months.
9. Documented left atrium (LA) thrombus on baseline/pre-procedure imaging.
10. LA antero posterior diameter > 50 mm
11. Any PV with a diameter ≥ 26 mm
12. Left Ventricular Ejection Fraction (LVEF) < 40%.
13. Contraindication to anticoagulation (e.g. heparin).
14. History of blood clotting or bleeding abnormalities.
15. Myocardial infarction within the past 2 months.
16. Documented thromboembolic event [including transient ischemic attack(TIA)] within the past 12 months.
17. Rheumatic Heart Disease.
18. Uncontrolled heart failure or New York Heart Association (NYHA) function class III or IV.
19. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months.
20. Unstable angina.
21. Acute illness or active systemic infection or sepsis.
22. Diagnosed atrial myxoma or interatrial baffle or patch.
23. Presence of implanted pacemaker or implantable cardioverter defibrillator (ICD).
24. Significant pulmonary disease, (e.g. restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
25. Significant congenital anomaly or medical problem that, in the opinion of the investigator, would preclude enrollment in this study.
26. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal), lactating, or who are of child bearing age and plan on becoming pregnant during the course of the clinical investigation.
27. Enrollment in an investigational study evaluating another device, biologic, or drug.
28. Has known pulmonary vein stenosis.
29. Presence of intramural thrombus, tumor or other abnormality that precludes vascular access, or manipulation of the catheter.
30. Presence of an Inferior Vena Cava (IVC) filter
31. Presence of a condition that precludes vascular access.
32. Life expectancy or other disease processes likely to limit survival to less than 12 months.
33. Presenting contra-indication for the devices (e.g. transthoracic echocardiography (TTE), CT, etc.) used in the study, as indicated in the respective instructions for use.
34. Categorized as a vulnerable population and requires special treatment with respect to safeguards of well-being

    Additional exclusion criteria for Neurological Assessment Evaluable (NAE) subjects:
35. Contraindication to use of contrast agents for MRI such as advanced renal disease, etc. (at PI discretion)
36. Presence of iron-containing metal fragments in the body
37. Unresolved pre-existing neurological deficit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Na Homolce Hospital, Prague, Czechia
- Italy (2):
  - Ospedale "F. Miulli", Bari
  - Centro Cardiologico Monzino, Milan
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - Bart's Health NHS Trust, London

REFERENCES:
- [Derived] Schilling R, Dhillon GS, Tondo C, Riva S, Grimaldi M, Quadrini F, Neuzil P, Chierchia GB, de Asmundis C, Abdelaal A, Vanderlinden L, Tan T, Ding WY, Gupta D, Reddy VY. Safety, effectiveness, and quality of life following pulmonary vein isolation with a multi-electrode radiofrequency balloon catheter in paroxysmal atrial fibrillation: 1-year outcomes from SHINE. Europace. 2021 Jun 7;23(6):851-860. doi: 10.1093/europace/euaa382. PMID 33450010

RESULTS

PARTICIPANT FLOW:
Groups:
- Roll-in Study Phase: RF Ablation: Roll-in study phase was to demonstrate the acute effectiveness of the multi-electrode RF balloon catheter in the absence of confounding evidence that reflects early stages of a medical device learning curve.
- Main Study Phase: RF Ablation: RF ablation was done using multi-electrode radiofrequency balloon catheter device (facilitate electrophysiological mapping of the heart and to transmit RF current to the target tissue) and multi-electrode circular diagnostic catheter device (recording and mapping of the atria of the heart with the carto system).
Period: Overall Study
Arm/Group | Roll-in Study Phase: RF Ablation | Main Study Phase: RF Ablation
Started | 8 | 90
Safety | 8 | 87
Completed | 8 | 87
Not Completed | 0 | 3
Not completed — Eligibility criteria not met | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Population included all enrolled participants who have undergone insertion of the study catheter.
Groups:
- Roll-in Study Phase: Radiofrequency (RF) Ablation: Roll-in study phase was to demonstrate the acute effectiveness of the multi-electrode RF balloon catheter in the absence of confounding evidence that reflects early stages of a medical device learning curve.
- Total: Total of all reporting groups
Arm/Group | Roll-in Study Phase: Radiofrequency (RF) Ablation | Main Study Phase: RF Ablation | Total
Number analyzed (Participants) | 8 | 87 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (6.90) | 60.2 (10.05) | 60.3 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 31 | 34
  Male | 5 | 56 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Onset Primary Adverse Events (PAEs): Death, Atrio-esophageal Fistula and Pulmonary Vein Stenosis
Description: A Primary AEs is an event which occurred within 90 days following initial ablation procedure. Primary AEs included: Death, atrio-esophageal fistula, and pulmonary vein stenosis.
Time Frame: Up to 90 days (post initial mapping and ablation procedure)
Population: The population analysis included the modified intent-to-treat (mITT) analysis set included all enrolled participants who met eligibility criteria, had undergone insertion of the study catheters and were followed-up for 90-days period for evaluation of PAEs.
Measure: Count of Participants; unit: Participants
Groups:
- Radiofrequency (RF) Ablation: RF ablation was done using multi-electrode radiofrequency balloon catheter device (facilitate electrophysiological mapping of the heart and to transmit RF current to the target tissue) and multi-electrode circular diagnostic catheter device (recording and mapping of the atria of the heart with the carto system).
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 84
Participants | 0

2. Primary Outcome: Number of Participants With Early Onset PAEs: Myocardial Infraction, Cardiac Tamponade/Perforation, Thromboembolism, Stroke/Cerebrovascular Accident, Transient Ischemic Attack, Phrenic Nerve Paralysis, and Major Vascular Access Complication/Bleeding
Description: A Primary AEs is an event which occurred within the first week (7 days of the initial mapping and ablation procedure) which included myocardial infraction (MI), cardiac tamponade (CT)/perforation, thromboembolism, stroke/cerebrovascular accident (CVA), Transient ischemic attack (TIA), phrenic nerve paralysis (PNP), and major vascular access complication (MVAC)/bleeding following initial ablation procedure.
Time Frame: Up to 7 days (post initial mapping and ablation procedure)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 84
Participants | 1

3. Primary Outcome: Percentage of Participants With Acute Procedural Success
Description: Acute procedural success is defined as confirmation of entrance block in treated pulmonary veins (PV) after adenosine and/or isoproterenol challenge (with or without the use of a focal catheter).
Time Frame: Day 1
Population: PP analysis set included participants who comply with the following criteria: a). were enrolled and met all eligibility criteria; b). had undergone RF ablation with study catheters; c) were treated for the study-related arrhythmia. Population included participants who had the adenosine/isoproterenol challenge.
Measure: Number; unit: Percentage of participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 82
Percentage of participants | 100

4. Secondary Outcome: Number of Participants With Individual PAE From Primary Composite
Description: A Primary AEs is an event which occurred within the first week (7 days of the initial mapping and ablation procedure) which included death, atrio-esophageal fistula (AE fistula) and pulmonary vein stenosis (PVST); and up to 90 days post procedure which included myocardial infraction (MI), cardiac tamponade (CT)/perforation, thromboembolism, stroke/cerebrovascular accident (CVA), Transient ischemic attack (TIA), phrenic nerve paralysis (PNP), and major vascular access complication (MVAC)/bleeding following initial ablation procedure.
Time Frame: Up to 7 days for MI, CT/perforation, thromboembolism, stroke/CVA, TIA, PNP and MVAC (initial mapping and ablation procedure) and up to 90 days for death, AE fistula, and PVST (post procedure)
Population: The population analysis included the mITT analysis set included all enrolled participants who met eligibility criteria, had undergone insertion of the study catheters and were followed-up for 90-days period for evaluation of PAEs. Here 'N' (number of participants analyzed) signifies the number of participants analyzed in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 84
Participants
  Death | 0
  Atrio-esophageal fistula | 0
  Myocardial infraction | 0
  Cardiac tamponade/perforation | 0
  Thromboembolism | 0
  Stroke/cerebrovascular accident (CVA) | 0
  Transient ischemic attack | 0
  Phrenic nerve paralysis | 0
  Pulmonary vein stenosis | 0
  Major vascular access complication/bleeding | 1

5. Secondary Outcome: Number of Participants With Serious Adverse Device Effects (SADEs)
Description: An adverse device effect is an adverse event related to the to the device and or the procedure of the investigational medical device. SADE is an adverse device effect that has resulted in any of the consequences characteristic of an SAE.
Time Frame: Up to 405 Days
Population: The safety population was defined to consist of all enrolled participants who have undergone insertion of the study catheter.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 87
Participants | 1

6. Secondary Outcome: Number of Participants With Serious Non-primary Adverse Events Within 7 Days (Early Onset), 8-30 Days (Peri-procedural) and Greater Than or Equal to (>=) 31 Days (Late Onset) of Initial Ablation Procedure
Description: Serious non-primary adverse event was defined as SAE that are not primary adverse events. Primary AEs included: Death, atrio-esophageal fistula, and pulmonary vein stenosis.
Time Frame: Within 7 Days (Early Onset), 8-30 Days (Peri-procedural) and >=31 Days (Late Onset) of Initial Ablation Procedure (Up to 405 Days)
Population: The safety population was defined to consist of all enrolled participants who have undergone insertion of the study catheter. Here 'n' (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 87
Participants
  0 - 7 Days | 0
  8 - 30 Days | 0
  >= 31 Days | 1

7. Secondary Outcome: Number of Participants With Non-serious Adverse Events
Description: An AE is any untoward medical occurrence in participants whether or not related to the investigational medical device.
Time Frame: Up to 405 Days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 87
Participants | 46

8. Secondary Outcome: Number of Participants With Pre-and Post-ablation Asymptomatic and Symptomatic Cerebral Emboli
Description: Number of participants with pre-and post-ablation asymptomatic and symptomatic cerebral emboli was reported.
Time Frame: Pre-procedure, at Discharge, 1 Month and at unscheduled visit (Up to 405 Days)
Population: Neurological Assessment Evaluable (NAE) Analysis set was a subset of the Per Protocol Population, consented and were eligible for the required neurological assessments, and had post-ablation MRI. Here 'n' (number analyzed) signifies participants with MRI done at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 31
Participants
  Pre-procedure | 0
  Discharge | 3
  1 Month: number analyzed (Participants) | 4
  1 Month | 0
  Unscheduled visit: number analyzed (Participants) | 1
  Unscheduled visit | 0

9. Secondary Outcome: Number of Participants With Symptomatic and Asymptomatic Cerebral Emboli
Description: Number of participants with symptomatic and asymptomatic cerebral emboli was reported
Time Frame: Up to 405 Days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 87
Participants
  Symptomatic | 0
  Asymptomatic | 4

10. Secondary Outcome: Number of Participants With New or Worsening Neurologic Deficits
Description: Number of participants with new or worsening neurologic deficits was reported.
Time Frame: Pre-procedure, discharge, 1 Month, 3 Month and 6 Month
Population: Neurological Assessment Evaluable (NAE) Analysis set was a subset of the Per Protocol Population, consented and were eligible for the required neurological assessments, and have post-ablation MRI. Here 'n' (number analyzed) signifies participants with neurological deficit at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 31
Participants
  Pre-procedure | 0
  Discharge | 1
  1 Month: number analyzed (Participants) | 4
  1 Month | 0
  3 Month: number analyzed (Participants) | 1
  3 Month | 0
  6 Month: number analyzed (Participants) | 1
  6 Month | 0

11. Secondary Outcome: Number of Participants With NIHSS Scores
Description: The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed to calculate a patient's total NIHSS score. The patient's total NIHSS score ranges from 0 (minimum) - 42 (maximum). Score 0 (no stroke symptoms); 1 - 4 (Minor stroke); 5-15 (Moderate stroke); 16-20 (Moderate to severe stroke); and 21-42 (Severe stroke).
Time Frame: Pre-procedure and at discharge (Up to 405 Days)
Population: NAE Analysis set was a subset of the Per Protocol Population, consent and are eligible for the required neurological assessments, and have post-ablation MRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 31
Participants
  Pre-procedure: NIHSS Score: 0 | 31
  Pre-procedure: NIHSS Score: 1-4 | 0
  Pre-procedure: NIHSS Score: 5-15 | 0
  Pre-procedure: NIHSS Score: 16-20 | 0
  Pre-procedure: NIHSS Score: 21-42 | 0
  Discharge: NIHSS Score: 0 | 31
  Discharge: NIHSS Score: 1-4 | 0
  Discharge: NIHSS Score: 5-15 | 0
  Discharge: NIHSS Score: 16-20 | 0
  Discharge: NIHSS Score: 21-42 | 0

12. Secondary Outcome: Number of Participants With MoCA Scores
Description: Montreal Cognitive Assessment (MoCA) is used for detecting cognitive impairment, the scores range from 0 to 30. A score of 26 or higher is considered normal, patients with mild cognitive impairment (MCI) were scored an average of 22 and patients with significant cognitive impairment (SCI) were scored an average of 16.
Time Frame: Up to 405 Days
Population: NAE Analysis set was a subset of the Per Protocol Population, consent and are eligible for the required neurological assessments, and have post-ablation MRI. Here 'n' (number analyzed) signifies participants analyzed at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 31
Participants
  Pre-procedure: 0-25 | 16
  Pre-procedure: 26-30 | 15
  1 Month: 0-25: number analyzed (Participants) | 30
  1 Month: 0-25 | 6
  1 Month: 26-30: number analyzed (Participants) | 30
  1 Month: 26-30 | 24
  3 Month: 0-25: number analyzed (Participants) | 2
  3 Month: 0-25 | 1
  3 Month: 26-30: number analyzed (Participants) | 2
  3 Month: 26-30 | 1
  6 Month: 0-25: number analyzed (Participants) | 1
  6 Month: 0-25 | 1
  6 Month: 26-30: number analyzed (Participants) | 1
  6 Month: 26-30 | 0

13. Secondary Outcome: Number of Participants With Hospitalization for Cardiovascular Events
Description: Hospitalization was defined as prolonged stay greater than or equal to (>=) 2 nights post index procedure or in-patient stay not concurrent with index procedure >= 1 calendar day. Hospitalization included cardiovascular events due to any cause post index procedure, regardless of protocol-defined serious/non-serious adverse events (AEs) or not. Hence this data was not contributed in serious Adverse events until met the AE definition.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 87
Participants
  0 - 7 Days | 2
  8 - 30 Days | 0
  >= 31 Days | 5

14. Secondary Outcome: Percentage of Participants With PVI Touch-up by Balloon and/or Focal Catheter Among All Targeted Veins and by Participants
Description: Percentage of participants with PVI touch-up by balloon and/or focal catheter among all targeted veins and by participants was reported. Most of the participants were ablated by Balloon catheter only while one participant was ablated with both Balloon and Focal catheters.
Time Frame: Up to 405 Days
Population: PP analysis set included participants who were enrolled and met all eligibility criteria; had undergone RF ablation with study catheters; and were treated for the study-related arrhythmia. Here 'n' (number analyzed) signifies number of pulmonary veins (PV) in all evaluable participants analyzed at specified category.
Measure: Number; unit: Percentage of participants
Units Other Than Participants: PV Veins
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 85
Number analyzed (PV Veins) | 327
Percentage of participants
  Balloon Catheter Ablation: Left Superior Pulmonary Vein (LSPV): number analyzed (Participants) | 84
  Balloon Catheter Ablation: Left Superior Pulmonary Vein (LSPV): number analyzed (PV Veins) | 76
  Balloon Catheter Ablation: Left Superior Pulmonary Vein (LSPV) | 100.0
  Balloon Catheter Ablation: Left Inferior Pulmonary Vein (LIPV): number analyzed (Participants) | 84
  Balloon Catheter Ablation: Left Inferior Pulmonary Vein (LIPV): number analyzed (PV Veins) | 75
  Balloon Catheter Ablation: Left Inferior Pulmonary Vein (LIPV) | 100.0
  Balloon Catheter Ablation: Right Superior Pulmonary Vein (RSPV): number analyzed (Participants) | 84
  Balloon Catheter Ablation: Right Superior Pulmonary Vein (RSPV): number analyzed (PV Veins) | 83
  Balloon Catheter Ablation: Right Superior Pulmonary Vein (RSPV) | 100.0
  Balloon Catheter Ablation: Right Inferior Pulmonary Vein (RIPV): number analyzed (Participants) | 84
  Balloon Catheter Ablation: Right Inferior Pulmonary Vein (RIPV): number analyzed (PV Veins) | 83
  Balloon Catheter Ablation: Right Inferior Pulmonary Vein (RIPV) | 98.8
  Balloon Catheter Ablation: Right Middle Pulmonary Vein (RMPV): number analyzed (Participants) | 84
  Balloon Catheter Ablation: Right Middle Pulmonary Vein (RMPV): number analyzed (PV Veins) | 1
  Balloon Catheter Ablation: Right Middle Pulmonary Vein (RMPV) | 100.0
  Balloon Catheter Ablation: Left Pulmonary Vein (LPV)-common: number analyzed (Participants) | 84
  Balloon Catheter Ablation: Left Pulmonary Vein (LPV)-common: number analyzed (PV Veins) | 9
  Balloon Catheter Ablation: Left Pulmonary Vein (LPV)-common | 100.0
  Balloon and Focal Catheter Ablation: LSPV: number analyzed (Participants) | 1
  Balloon and Focal Catheter Ablation: LSPV: number analyzed (PV Veins) | 76
  Balloon and Focal Catheter Ablation: LSPV | 0.0
  Balloon and Focal Catheter Ablation: LIPV: number analyzed (Participants) | 1
  Balloon and Focal Catheter Ablation: LIPV: number analyzed (PV Veins) | 75
  Balloon and Focal Catheter Ablation: LIPV | 0.0
  Balloon and Focal Catheter Ablation: RSPV: number analyzed (Participants) | 1
  Balloon and Focal Catheter Ablation: RSPV: number analyzed (PV Veins) | 83
  Balloon and Focal Catheter Ablation: RSPV | 0.0
  Balloon and Focal Catheter Ablation: RIPV: number analyzed (Participants) | 1
  Balloon and Focal Catheter Ablation: RIPV: number analyzed (PV Veins) | 83
  Balloon and Focal Catheter Ablation: RIPV | 1
  Balloon and Focal Catheter Ablation: RMPV: number analyzed (Participants) | 1
  Balloon and Focal Catheter Ablation: RMPV: number analyzed (PV Veins) | 1
  Balloon and Focal Catheter Ablation: RMPV | 0.0
  Balloon and Focal Catheter Ablation: LPV-common: number analyzed (Participants) | 1
  Balloon and Focal Catheter Ablation: LPV-common: number analyzed (PV Veins) | 9
  Balloon and Focal Catheter Ablation: LPV-common | 0.0

15. Secondary Outcome: Percentage of Participants With Use of Focal Catheter Ablation for Non-PV Triggers
Description: Percentage of participants with use of focal catheter ablation for non-PV triggers was reported.
Time Frame: Up to 405 Days
Population: PP analysis set included participants who comply with the following criteria: a). were enrolled and met all eligibility criteria; b). had undergone RF ablation with study catheters; c) were treated for the study-related arrhythmia.
Measure: Number; unit: Percentage of participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 85
Percentage of participants | 3.5

16. Secondary Outcome: Percentage of Participants With Freedom From Documented Atrial Fibrillation (AF), Atrial Tachycardia (AT), or Atypical (Left Side) Atrial Flutter (AFL) Episodes or Documented Symptomatic AF/AT/AFL
Description: Percentage of participants with six-month arrythmia recurrence [defined as freedom from documented symptomatic or asymptomatic atrial fibrillation (AF), atrial tachycardia (AT), or atypical (left side) atrial flutter (AFL) episodes (episodes >30 seconds on arrhythmia monitoring device from Day 91 to 180 post the index procedure)] was reported.
Time Frame: Up to 6 Months
Population: PP analysis set included participants who comply with the following criteria: a). were enrolled and met all eligibility criteria; b). had undergone RF ablation with study catheters; c) were treated for the study-related arrhythmia. Here 'N' (number of participants analyzed) signifies the number of participants analyzed in this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 84
Percentage of participants
  Documented AF/AT/AFL | 76.2
  Documented Symptomatic AF/AT/AFL | 81.0

17. Secondary Outcome: Percentage of Participants With Freedom From Documented, AF, AT, or Atypical (Left Side) AFL Episodes or Documented Symptomatic AF/AT/AFL
Description: Twelve-month Arrythmia recurrence is defined as a documented symptomatic or asymptomatic episode >30 seconds on an arrhythmia monitoring device between day 91 to 365 post the index procedure.
Time Frame: Up to 12 Months
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | Radiofrequency (RF) Ablation
Number analyzed (Participants) | 79
Percentage of participants
  Documented AF/AT/AFL | 65.8
  Documented Symptomatic AF/AT/AFL | 72.2

ADVERSE EVENTS:
Time Frame: Up to 405 Days
Description: The safety population included all participants who have undergone insertion of the study catheter.
Arm/Group | Roll-in Study Phase: RF Ablation | Main Study Phase: RF Ablation
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/87
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/87
Other Adverse Events (participants affected / at risk) | 0/8 | 0/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roll-in Study Phase: RF Ablation (N=8) | Main Study Phase: RF Ablation (N=87)
Major Vascular Access Complication/ Bleeding (Cardiac disorders) | 0 | 1
ST-elevation myocardial infarction (Cardiac disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03437733/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03437733/SAP_001.pdf